CLINICAL TRIAL: NCT03716609
Title: Effects of Magnesium Supplementation on Hemodynamic Parameters and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Wen-Harn Pan, Distinguished Research Fellow, Academia Sinica, Taiwan
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: AS-IRB-BM-18037
Record Dates: First submitted 2018-10-22; First posted 2018-10-23 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Function
MeSH Terms: interventions — magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium supplement group (Experimental): Subjects receive citrate acid drinks with additional magnesium citrate (300mg magnesium)
  Interventions: Dietary Supplement: Magnesium Citrate; Other: Food grade citrate acid; Other: Splenda(Sucralose)
- placebo group (Placebo Comparator): Subjects receive citrate acid drinks without additional magnesium
  Interventions: Other: Food grade citrate acid; Other: Splenda(Sucralose)

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate — Pure Magnesium citrate powder 2.07 gram from NOW FOODS (Bloomingdale, IL, USA)
  Arms: Magnesium supplement group
Other: Food grade citrate acid — Food grade citrate acid 0.1 gram from San Fu Chemical Co., Ltd (Taipei, Taiwan)
Other: Splenda(Sucralose) — Splenda 1.0 gram from Splenda(Carmel, Indiana, USA)

SUMMARY:
Using a double-blind randomized controlled trial design, this study intends to evaluate the short-term effect of magnesium citrate on cognitive functions and hemodynamic parameters in MCI elders, including Montreal Cognitive Assessment, working memory test-digit span test, carotid artery flow velocity, ankle-brachial blood pressure ratio, and urinary magnesium.

DETAILED DESCRIPTION:
Dementia is an important geriatric syndrome. The prevalence of dementia increases with age. According to the data of the Taiwan Alzheimer Disease Association, one out of 13 elderly people over 65 and one out of 5 elderly over 80 had dementia. Almost 20% of the elderly people have the mild cognitive impairment (MCI), an intermediate stage between normal cognition and dementia. The results from the Nutrition and Health Survey in Taiwan (NAHSIT), 2013-2016 found that magnesium average intake was much lower than the daily recommended intake level in MCI elders over 65. Since magnesium, an abundant essential mineral in human body plays important roles in energy provision, anti-inflammation, and preventing post-stroke NMDA toxicity; our previous study trialed and showed that a moderate level of daily magnesium supplementation could improve stroke recovery for discharged stroke patients in a 6-month clinical trial. Due to its effect on neuroprotection, this study intends to evaluate the short-term effect of magnesium supplement at a DRI level on cognitive function and on certain hemodynamic parameters.

MCI participants aged 60 and over are eligible for recruitment. The Mini-Mental State Examination (MMSE) will be used to determine the MCI status. A score of 25 or lower is indicative of cognitive impairment. The exclusion criteria include: regularly taking magnesium supplements, having a severe illness (e.g. cancer), bed-ridden, inability to speak, with visual or hearing impairment, and living in elderly homes.

The investigators designed a double-blind randomized controlled trial. Participants will be divided into magnesium intervention group and placebo group. Participants of the placebo group will receive 30cc solution containing 100 mg of citrate acid and flavored by 1g of Splenda. The magnesium citrate pure powder from NOW FOODS containing 300mg magnesium will be dissolved in 30cc of the above solution.

Before and after two hours of intervention, participants will be interviewed and assessed for the following: questionnaires, cognitive function, carotid artery flow velocity, ankle-brachial blood pressure ratio, and urinary magnesium. Questionnaires include Montreal Cognitive Assessment (MoCA) and working memory test - digit span test. Philips iE33 Ultrasound System and OMRON Non-invasive Vascular Screening Device VP1000 plus will be used to measure carotid artery flow velocity and ankle-brachial blood pressure ratio.

This intervention will be carried out after the informed consent form is signed, roughly from 8 AM in the morning to 12:30 PM. Participants have to take their breakfast before the trial and allowed to eat lunch after the process finishes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mild cognitive impairment (Mini-Metal State Examination < 26 points)
* Participants signing the informed consent form

Exclusion Criteria:

* Participants regularly taking magnesium supplements
* Participants who had severe illness (e.g. cancer, ridden bed)
* Participants unable to speak, with visual disorder and hearing impairment)
* Participants hospitalized who live in elderly homes

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
End-diastolic velocity | Two hours from intervention to follow-up measurement
  End-diastolic velocity of internal carotid artery

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Harn Pan, Ph.D., Principal Investigator — Institute of Biomedical Sciences, Academia Sinica
Locations (1):
- Academia Sinica, Taipei, Taiwan